CLINICAL TRIAL: NCT02715206
Title: Adaptation Processes in School-based Substance Abuse Prevention
Acronym: kiR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Michael L. Hecht, Distinguished Professor of Communication Arts and Sciences, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA021670 (NIH)
Record Dates: First submitted 2016-02-25; First posted 2016-03-22 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Substance Abuse Problem
Keywords: rural adolescents, substance use, prevention, adaptation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Experimental): middle schools not receiving keepin' it REAL; continue their own programs if any.
  Interventions: Behavioral: control
- keepin' it REAL classic (Experimental): middle schools will implement keepin' it REAL classic drug prevention curriculum
  Interventions: Behavioral: keepin' it REAL classic
- keepin' it REAL rural (Experimental): middle schools will implement the keepin' it REAL rural curriculum
  Interventions: Behavioral: keepin' it REAL rural

INTERVENTIONS:
Behavioral: keepin' it REAL classic — keepin' it REAL consists of 10 classroom lessons implemented in 7th grade and 4 booster sessions implemented in 8th grade by the classroom teacher following training
  Arms: keepin' it REAL classic
Behavioral: keepin' it REAL rural — keepin' it REAL rural drug prevention curriculum consists for 10 lessons taught in 7th grade and 4 booster sessions taught in 8th grade.
  Arms: keepin' it REAL rural
Behavioral: control — control group continues to teach whatever prevention curriculum they were using prior to study
  Arms: Control

SUMMARY:
The purpose of this study is to determine if a new substance use prevention curriculum for rural middle schools is effective in reducing substance use and to study how prevention curriculum get implemented by teachers.

DETAILED DESCRIPTION:
The goals of the proposed study are to conduct an effectiveness trial of the keepin' it REAL (refuse, explain, avoid, leave) middle school substance use prevention curriculum among a new target audience in rural Pennsylvania and Ohio, describe how teachers adapt the curriculum when they present it, and develop, implement, and evaluate a Pennsylvania/Ohio-version of the curriculum to test whether an evidence-based universal curriculum can be improved by adapting it to local cultures. keepin' it REAL is recognized as a "model program" by SAMHSA's (Substance Abuse and Mental Health Services Administration's) National Registry of Effective programs and is one of the few that are multicultural. The study will evaluate the effectiveness of the original curriculum, grounded in the cultures of the southwest and compare that to a new version, "re-grounded" in the rural culture of Pennsylvania and Ohio, while studying how teachers adapt both versions. This proposal responds to NIDA (National Institute on Drug Abuse) PA-05-118 (Program Announcement), Drug Abuse Prevention Intervention Research that calls for investigations addressing, "1) the development of novel drug abuse prevention approaches; 2) the efficacy and effectiveness of newly developed and/or modified prevention programs; 3) the processes associated with the selection, adoption, adaptation, implementation, sustainability, and financing of empirically validated interventions." This proposal addresses all three points.

A randomized control trial will be conducted in middle schools to accomplish these goals. First, formative research will be conducted to develop a rural Pennsylvania/Ohio-version of the curriculum. Second, 39 rural schools will be randomly assigned to one of three conditions: teacher adaptation in which the original keepin' it REAL curriculum is implemented; researcher adaptation in which a new Pennsylvania-version of the curriculum is implemented, and a control group. We hypothesized the participation in either form of the curriculum will reduce drug use and that the researcher adaptation will produce better outcomes and less teacher adaptation than the teacher adaptation. A pretest will be administered followed by post-tests in 7-9th grades. Adaptation and fidelity will be measured in 3 ways: teachers completing a Program Quality and Adaptation online measure after each lesson, videotaped lessons, and attendance. The major hypothesis tests will be conducted using variants of the general linear model, taking into account the multilevel structure of the data, test of a mediation model, and growth modeling.

ELIGIBILITY:
Inclusion Criteria:

- all 7th grade students in implementation middle

Exclusion Criteria:

* lack of parental consent
* lack of student assent

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2827 (Actual)
Dates: Start 2006-07; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Recent use of alcohol | 30 days
  Self report measure of recent use of alcohol
Recent use of tobacco | 30 days
  Self report measure
Recent use of marijuana | 30 days
  Self report

SECONDARY OUTCOMES:
Perceptions of number of peers using drugs | 2 years
  Self report
Perception of self efficacy resisting drug offers | 2 years
  Self report measure

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Hecht, PhD, Principal Investigator — The Pennsylvania State University
Locations (2):
- United States (2):
  - The Ohio State University, Columbus, Ohio
  - The Pennsylvania State University, University Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Graham JW, Pettigrew J, Miller-Day M, Krieger JL, Zhou J, Hecht ML. Random assignment of schools to groups in the drug resistance strategies rural project: some new methodological twists. Prev Sci. 2014 Aug;15(4):516-25. doi: 10.1007/s11121-013-0403-9. PMID 23722619
- [Background] Shin Y, Miller-Day M, Pettigrew J, Hecht ML, Krieger JL. Typology of delivery quality: latent profile analysis of teacher engagement and delivery techniques in a school-based prevention intervention, keepin' it REAL curriculum. Health Educ Res. 2014 Dec;29(6):897-905. doi: 10.1093/her/cyu061. Epub 2014 Sep 30. PMID 25274721
- [Background] Choi HJ, Krieger JL, Hecht ML. Reconceptualizing efficacy in substance use prevention research: refusal response efficacy and drug resistance self-efficacy in adolescent substance use. Health Commun. 2013;28(1):40-52. doi: 10.1080/10410236.2012.720245. PMID 23330857
- [Background] Krieger JL, Coveleski S, Hecht ML, Miller-Day M, Graham JW, Pettigrew J, Kootsikas A. From kids, through kids, to kids: examining the social influence strategies used by adolescents to promote prevention among peers. Health Commun. 2013;28(7):683-95. doi: 10.1080/10410236.2012.762827. Epub 2013 Aug 27. PMID 23980520
- [Background] Colby M, Hecht ML, Miller-Day M, Krieger JL, Syvertsen AK, Graham JW, Pettigrew J. Adapting school-based substance use prevention curriculum through cultural grounding: a review and exemplar of adaptation processes for rural schools. Am J Community Psychol. 2013 Mar;51(1-2):190-205. doi: 10.1007/s10464-012-9524-8. PMID 22961604
- [Background] Hopfer S, Hecht ML, Lanza ST, Tan X, Xu S. Preadolescent drug use resistance skill profiles, substance use, and substance use prevention. J Prim Prev. 2013 Dec;34(6):395-404. doi: 10.1007/s10935-013-0325-0. PMID 23990398
- [Background] Miller-Day M, Pettigrew J, Hecht ML, Shin Y, Graham J, Krieger J. How prevention curricula are taught under real-world conditions: Types of and reasons for teacher curriculum adaptations. Health Educ (Lond). 2013;113(4):324-344. doi: 10.1108/09654281311329259. PMID 26290626
- [Background] Moreland JJ, Raup-Krieger JL, Hecht ML, Miller-Day MM. The conceptualization and communication of risk among rural appalachian adolescents. J Health Commun. 2013;18(6):668-85. doi: 10.1080/10810730.2012.743620. Epub 2013 Feb 28. PMID 23448190
- [Background] Pettigrew J, Miller-Day M, Shin Y, Hecht ML, Krieger JL, Graham JW. Describing teacher-student interactions: a qualitative assessment of teacher implementation of the 7th grade keepin' it REAL substance use intervention. Am J Community Psychol. 2013 Mar;51(1-2):43-56. doi: 10.1007/s10464-012-9539-1. PMID 22739791
- [Background] Pettigrew J, Miller-Day M, Krieger J, Hecht ML. The Rural Context of Illicit Substance Offers: A Study of Appalachian Rural Adolescents. J Adolesc Res. 2012 Jul;27(4):523-550. doi: 10.1177/0743558411432639. PMID 25620838
- [Background] Pettigrew J, Miller-Day M, Krieger J, Hecht ML. Alcohol and Other Drug Resistance Strategies Employed by Rural Adolescents. J Appl Commun Res. 2011;39(2):103-122. doi: 10.1080/00909882.2011.556139. PMID 21552345
- [Result] Miller-Day M, Hecht ML, Krieger JL, Pettigrew J, Shin Y, Graham J. Teacher Narratives and Student Engagement: Testing Narrative Engagement Theory in Drug Prevention Education. J Lang Soc Psychol. 2015 Dec 1;34(6):604-620. doi: 10.1177/0261927X15586429. Epub 2015 May 14. PMID 26690668
- [Result] Pettigrew J, Graham JW, Miller-Day M, Hecht ML, Krieger JL, Shin YJ. Erratum to: Adherence and Delivery: Implementation Quality and Program Outcomes for the Seventh-Grade keepin' it REAL Program. Prev Sci. 2015 Jan;16(1):100. doi: 10.1007/s11121-014-0506-y. No abstract available. PMID 25274060